CLINICAL TRIAL: NCT04887948
Title: A PHASE 3, RANDOMIZED, DOUBLE BLIND TRIAL TO DESCRIBE THE SAFETY AND IMMUNOGENICITY OF 20 VALENT PNEUMOCOCCAL CONJUGATE VACCINE WHEN COADMINISTERED WITH A BOOSTER DOSE OF BNT162b2 IN ADULTS 65 YEARS OF AGE AND OLDER
Brief Title: Safety and Immunogenicity Study of 20vPnC When Coadministered With a Booster Dose of BNT162b2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B7471026
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Results first posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Pneumococcal Disease; COVID-19; SARS-CoV-2 Infection
MeSH Terms: conditions — Pneumococcal Infections; COVID-19 | interventions — BNT162 Vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Coadministration Group (Experimental): Participants receive an injection of pneumococcal vaccine (20vPnC) and of COVID-19 vaccine (BNT162b2) at the same visit.
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine (20vPnC); Biological: BNT162b2
- 20vPnC-only Group (Active Comparator): Participants receive an injection of pneumococcal vaccine (20vPnC) and of saline at the same visit.
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine (20vPnC); Other: Saline
- BNT162b2-only Group (Active Comparator): Participants receive an injection of COVID-19 vaccine (BNT162b2) and of saline at the same visit.
  Interventions: Biological: BNT162b2; Other: Saline

INTERVENTIONS:
Biological: 20-valent pneumococcal conjugate vaccine (20vPnC) — 20-valent pneumococcal conjugate vaccine (20vPnC)
  Arms: 20vPnC-only Group; Coadministration Group
Biological: BNT162b2 — RNA-based SARS-CoV-2 vaccine (BNT162b2)
  Arms: BNT162b2-only Group; Coadministration Group
Other: Saline — Normal saline for injection
  Arms: 20vPnC-only Group; BNT162b2-only Group

SUMMARY:
Study of the safety and immunogenicity of 20vPnC and a booster dose of BNT162b2 administered at the same visit or each vaccine given alone

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥65 years of age at the time of consent
* Participating or participated in Study C4591001, received 2 doses of 30 µg BNT162b2 with the second dose given ≥6 months prior to the first vaccination in this study, and have not received a third dose of BNT162b2
* Adults determined by clinical assessment, including medical history and clinical judgement, to be eligible for the study, including adults with preexisting stable disease
* Adults who have no history of ever receiving a pneumococcal vaccine, or received a licensed pneumococcal vaccination ≥12 months prior to the first vaccination in this study

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis)
* Serious chronic disorder that in the investigator's opinion would make the participant inappropriate for entry into the study
* Previous clinical or microbiological diagnosis of COVID-19
* Previous vaccination with any investigational pneumococcal vaccine, or planned receipt of any licensed or investigational pneumococcal vaccine through study participation
* Previous vaccination with any coronavirus vaccine, other than those received in Study C4591001
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 570 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- United States (27):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Alliance for Multispecialty Research, LLC, Coral Gables, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Solaris Clinical Research, Meridian, Idaho
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Clinical Research Professionals, Chesterfield, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Meridian Clinical Research, LLC, Endwell, New York
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Aventiv Research Inc, Columbus, Ohio
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Memphis, Tennessee
  - Benchmark Research, Austin, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - Martins Diagnostic Clinic, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Wenatchee Valley Hospital, Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Fitz-Patrick D, Young M, Yacisin K, McElwee K, Belanger T, Belanger K, Peng Y, Lee DY, Gruber WC, Scott DA, Watson W. Randomized trial to evaluate the safety, tolerability, and immunogenicity of a booster (third dose) of BNT162b2 COVID-19 vaccine coadministered with 20-valent pneumococcal conjugate vaccine in adults >/=65 years old. Vaccine. 2023 Jun 23;41(28):4190-4198. doi: 10.1016/j.vaccine.2023.05.002. Epub 2023 May 8. PMID 37244809
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471026

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants who received 2 doses of ribonucleic acid (RNA)-based COVID-19 vaccine (BNT162b2) at least 6 months previously in study C4591001 (NCT04368728) were stratified by prior pneumococcal vaccine status (no previous pneumococcal vaccine [naïve] or receipt of at least 1 dose of a pneumococcal vaccine [experienced]) and randomized to 1 of the 3 vaccine groups in this study.
Pre-assignment Details: A total of 570 participants were enrolled in the study and randomized to a study treatment.
Groups:
- Coadministration Group: 20vPnC+BNT162b2: On Day 1, participants were randomized to receive a single dose of 0.5 milliliter (mL) 20-valent pneumococcal conjugate vaccine (20vPnC) intramuscularly into the right deltoid and a single dose of 0.3 mL booster dose of BNT162b2 intramuscularly into the left deltoid. Participants were followed up for 6 months after vaccination.
- 20vPnC Only Group: 20vPnC+Saline: On Day 1, participants were randomized to receive a single dose of 0.5 mL 20vPnC intramuscularly into the right deltoid and a single dose of 0.3 mL saline intramuscularly into the left deltoid. Participants were followed up for 6 months after vaccination.
- BNT162b2 Only Group: BNT162b2+Saline: On Day 1, participants were randomized to receive a single dose of 0.5 mL saline intramuscularly into the right deltoid and a single dose of 0.3 mL booster dose of BNT162b2 intramuscularly into the left deltoid. Participants were followed up for 6 months after vaccination.
Period: Overall Study
Arm/Group | Coadministration Group: 20vPnC+BNT162b2 | 20vPnC Only Group: 20vPnC+Saline | BNT162b2 Only Group: BNT162b2+Saline
Started | 190 | 191 | 189
Vaccinated | 187 | 187 | 185
Completed | 184 | 177 | 182
Not Completed | 6 | 14 | 7
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 3
Not completed — Physician Decision | 0 | 4 | 1
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 6 | 1
Not completed — No longer met eligibility criteria | 1 | 2 | 1
Not completed — Other | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of the study intervention and had safety follow-up after vaccination.
Groups:
- Coadministration Group: 20vPnC+BNT162b2: On Day 1, participants were randomized to receive a single dose of 0.5 mL 20vPnC intramuscularly into the right deltoid and a single dose of 0.3 mL booster dose of BNT162b2 intramuscularly into the left deltoid. Participants were followed up for 6 months after vaccination.
- Total: Total of all reporting groups
Arm/Group | Coadministration Group: 20vPnC+BNT162b2 | 20vPnC Only Group: 20vPnC+Saline | BNT162b2 Only Group: BNT162b2+Saline | Total
Number analyzed (Participants) | 187 | 187 | 185 | 559
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.0 (4.22) | 71.8 (4.94) | 71.8 (4.95) | 71.5 (4.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 75 | 77 | 241
  Male | 98 | 112 | 108 | 318
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 26 | 25 | 79
  Not Hispanic or Latino | 159 | 161 | 160 | 480
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 10 | 5 | 9 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 7 | 10 | 25
  White | 164 | 172 | 165 | 501
  More than one race | 4 | 2 | 0 | 6
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions at Each Injection Site Within 10 Days After Vaccination
Description: Local reactions included pain at injection site, redness and swelling and were recorded by participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm) and graded as mild: greater than (>) 2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm and severe: >10.0 cm. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity and severe: prevented daily activity. Percentage of participants with local reactions at each injection site within 10 days after vaccination and the associated 2-sided 95% confidence interval (CI) based on the Clopper and Pearson method was presented.
Time Frame: Within 10 days after vaccination
Population: Safety population included all participants who received at least 1 dose of the study intervention and had safety follow-up after vaccination. Here, "Overall Number of Participants Analyzed" signifies number of participants with any e-diary data reported after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Coadministration Group (20vPnC+BNT162b2): 20vPnC Vaccination Site; 20vPnC Only Group (20vPnC+Saline): 20vPnC Vaccination Site: On Day 1, participants were randomized to receive a single dose of 0.5 mL 20vPnC intramuscularly into the right deltoid. Participants were followed up for 6 months after vaccination.
- Coadministration Group (20vPnC+BNT162b2): BNT162b2 Vaccination Site; BNT162b2 Only Group (BNT162b2+Saline): BNT162b2 Vaccination Site: On Day 1, participants were randomized to receive a single dose of 0.3 mL booster dose of BNT162b2 intramuscularly into the left deltoid. Participants were followed up for 6 months after vaccination.
- 20vPnC Only Group (20vPnC+Saline): Saline Vaccination Site: On Day 1, participants were randomized to receive a single dose of 0.3 mL saline intramuscularly into the left deltoid. Participants were followed up for 6 months after vaccination.
- BNT162b2 Only Group (BNT162b2+Saline): Saline Vaccination Site: On Day 1, participants were randomized to receive a single dose of 0.5 mL saline intramuscularly into the right deltoid. Participants were followed up for 6 months after vaccination.
Arm/Group | Coadministration Group (20vPnC+BNT162b2): 20vPnC Vaccination Site | Coadministration Group (20vPnC+BNT162b2): BNT162b2 Vaccination Site | 20vPnC Only Group (20vPnC+Saline): 20vPnC Vaccination Site | 20vPnC Only Group (20vPnC+Saline): Saline Vaccination Site | BNT162b2 Only Group (BNT162b2+Saline): BNT162b2 Vaccination Site | BNT162b2 Only Group (BNT162b2+Saline): Saline Vaccination Site
Number analyzed (Participants) | 185 | 185 | 186 | 186 | 185 | 185
Percentage of participants
  Redness: Any | 8.6 [5.0 to 13.7] | 9.7 [5.9 to 14.9] | 8.1 [4.6 to 13.0] | 0.0 [0.0 to 2.0] | 9.7 [5.9 to 14.9] | 2.7 [0.9 to 6.2]
  Redness: Mild | 5.9 [3.0 to 10.4] | 5.9 [3.0 to 10.4] | 4.3 [1.9 to 8.3] | 0.0 [0.0 to 2.0] | 6.5 [3.4 to 11.1] | 2.2 [0.6 to 5.4]
  Redness: Moderate | 2.7 [0.9 to 6.2] | 3.2 [1.2 to 6.9] | 3.2 [1.2 to 6.9] | 0.0 [0.0 to 2.0] | 2.7 [0.9 to 6.2] | 0.5 [0.0 to 3.0]
  Redness: Severe | 0.0 [0.0 to 2.0] | 0.5 [0.0 to 3.0] | 0.5 [0.0 to 3.0] | 0.0 [0.0 to 2.0] | 0.5 [0.0 to 3.0] | 0.0 [0.0 to 2.0]
  Swelling: Any | 8.1 [4.6 to 13.0] | 9.7 [5.9 to 14.9] | 8.6 [5.0 to 13.6] | 0.0 [0.0 to 2.0] | 11.4 [7.2 to 16.8] | 1.1 [0.1 to 3.9]
  Swelling: Mild | 5.4 [2.6 to 9.7] | 5.9 [3.0 to 10.4] | 5.4 [2.6 to 9.7] | 0.0 [0.0 to 2.0] | 6.5 [3.4 to 11.1] | 0.0 [0.0 to 2.0]
  Swelling: Moderate | 2.7 [0.9 to 6.2] | 3.8 [1.5 to 7.6] | 3.2 [1.2 to 6.9] | 0.0 [0.0 to 2.0] | 4.9 [2.2 to 9.0] | 1.1 [0.1 to 3.9]
  Swelling: Severe | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Pain at injection site: Any | 73.0 [66.0 to 79.2] | 72.4 [65.4 to 78.7] | 60.2 [52.8 to 67.3] | 9.7 [5.8 to 14.9] | 67.6 [60.3 to 74.3] | 16.8 [11.7 to 22.9]
  Pain at injection site: Mild | 55.1 [47.7 to 62.4] | 56.8 [49.3 to 64.0] | 52.2 [44.7 to 59.5] | 9.7 [5.8 to 14.9] | 50.3 [42.8 to 57.7] | 16.2 [11.2 to 22.3]
  Pain at injection site: Moderate | 17.8 [12.6 to 24.1] | 15.7 [10.8 to 21.7] | 7.0 [3.8 to 11.7] | 0.0 [0.0 to 2.0] | 17.3 [12.1 to 23.5] | 0.5 [0.0 to 3.0]
  Pain at injection site: Severe | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0] | 1.1 [0.1 to 3.8] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]

2. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination
Description: Systemic events including fever, fatigue, headache, chills, muscle pain and joint pain were recorded by participants using an e-diary. Fever was defined as temperature >=38.0 degree Celsius (C) and categorized as >=38.0 to 38.4 degree C, >38.4 to 38.9 degree C, >38.9 to 40.0 degree C and >40.0 degree C. Fatigue, headache, chills, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Percentage of participants with systemic events within 7 days after vaccination and the associated 2-sided 95% CI based on the Clopper and Pearson method was presented.
Time Frame: Within 7 days after vaccination
Population: Safety population included all participants who received at least 1 dose of the study intervention and had safety follow-up after vaccination. Here, "Overall Number of Participants Analyzed" (N) signifies number of participants with any e-diary data reported after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Coadministration Group: 20vPnC+BNT162b2 | 20vPnC Only Group: 20vPnC+Saline | BNT162b2 Only Group: BNT162b2+Saline
Number analyzed (Participants) | 185 | 186 | 185
Percentage of participants
  Fever: >=38.0 degree C | 13.0 [8.5 to 18.7] | 1.1 [0.1 to 3.8] | 8.6 [5.0 to 13.7]
  Fever: >=38.0 degree C to 38.4 degree C | 7.0 [3.8 to 11.7] | 0.5 [0.0 to 3.0] | 2.7 [0.9 to 6.2]
  Fever: >38.4 degree C to 38.9 degree C | 5.4 [2.6 to 9.7] | 0.5 [0.0 to 3.0] | 4.9 [2.2 to 9.0]
  Fever: >38.9 degree C to 40.0 degree C | 0.5 [0.0 to 3.0] | 0.0 [0.0 to 2.0] | 1.1 [0.1 to 3.9]
  Fever: >40.0 degree C | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Fatigue: Any | 54.1 [46.6 to 61.4] | 36.0 [29.1 to 43.4] | 54.6 [47.1 to 61.9]
  Fatigue: Mild | 17.8 [12.6 to 24.1] | 23.7 [17.7 to 30.4] | 27.0 [20.8 to 34.0]
  Fatigue: Moderate | 33.0 [26.3 to 40.3] | 12.4 [8.0 to 18.0] | 24.9 [18.8 to 31.7]
  Fatigue: Severe | 3.2 [1.2 to 6.9] | 0.0 [0.0 to 2.0] | 2.7 [0.9 to 6.2]
  Headache: Any | 30.3 [23.7 to 37.4] | 17.2 [12.1 to 23.4] | 33.0 [26.3 to 40.3]
  Headache: Mild | 17.8 [12.6 to 24.1] | 14.5 [9.8 to 20.4] | 24.9 [18.8 to 31.7]
  Headache: Moderate | 11.9 [7.6 to 17.4] | 2.7 [0.9 to 6.2] | 7.6 [4.2 to 12.4]
  Headache: Severe | 0.5 [0.0 to 3.0] | 0.0 [0.0 to 2.0] | 0.5 [0.0 to 3.0]
  Chills: Any | 26.5 [20.3 to 33.5] | 7.0 [3.8 to 11.7] | 22.2 [16.4 to 28.8]
  Chills: Mild | 18.4 [13.1 to 24.7] | 5.9 [3.0 to 10.3] | 12.4 [8.0 to 18.1]
  Chills: Moderate | 6.5 [3.4 to 11.1] | 1.1 [0.1 to 3.8] | 7.6 [4.2 to 12.4]
  Chills: Severe | 1.6 [0.3 to 4.7] | 0.0 [0.0 to 2.0] | 2.2 [0.6 to 5.4]
  Muscle pain: Any | 32.4 [25.7 to 39.7] | 14.5 [9.8 to 20.4] | 31.9 [25.2 to 39.1]
  Muscle pain: Mild | 17.3 [12.1 to 23.5] | 10.2 [6.3 to 15.5] | 15.7 [10.8 to 21.7]
  Muscle pain: Moderate | 14.1 [9.4 to 19.9] | 4.3 [1.9 to 8.3] | 15.1 [10.3 to 21.1]
  Muscle pain: Severe | 1.1 [0.1 to 3.9] | 0.0 [0.0 to 2.0] | 1.1 [0.1 to 3.9]
  Joint pain: Any | 26.5 [20.3 to 33.5] | 9.1 [5.4 to 14.2] | 24.9 [18.8 to 31.7]
  Joint pain: Mild | 15.1 [10.3 to 21.1] | 5.4 [2.6 to 9.7] | 15.1 [10.3 to 21.1]
  Joint pain: Moderate | 11.4 [7.2 to 16.8] | 3.8 [1.5 to 7.6] | 9.7 [5.9 to 14.9]
  Joint pain: Severe | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Vaccination
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants with AEs and the associated 2-sided 95% CI based on the Clopper and Pearson method was presented. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From day of vaccination (Day 1) up to 1 month after vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Coadministration Group: 20vPnC+BNT162b2 | 20vPnC Only Group: 20vPnC+Saline | BNT162b2 Only Group: BNT162b2+Saline
Number analyzed (Participants) | 187 | 187 | 185
Percentage of participants | 5.3 [2.6 to 9.6] | 4.3 [1.9 to 8.3] | 6.5 [3.4 to 11.1]

4. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Within 6 Months After Vaccination
Description: A SAE was defined as any untoward medical occurrence that, at any dose, resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect; was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic or that was considered to be an important medical event. Percentage of participants with SAEs and the associated 2-sided 95% CI based on the Clopper and Pearson method was presented.
Time Frame: From day of vaccination (Day 1) up to 6 months after vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Coadministration Group: 20vPnC+BNT162b2 | 20vPnC Only Group: 20vPnC+Saline | BNT162b2 Only Group: BNT162b2+Saline
Number analyzed (Participants) | 187 | 187 | 185
Percentage of participants | 0.5 [0.0 to 2.9] | 1.1 [0.1 to 3.8] | 2.7 [0.9 to 6.2]

5. Secondary Outcome: Geometric Mean Titers (GMTs) of Pneumococcal Serotype-Specific Opsonophagocytic Activity (OPA) at 1 Month After Vaccination With 20vPnC
Description: OPA titers were measured from serum samples for 20vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F,8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, and 33F. GMTs and 2-sided CIs were calculated by exponentiating the mean logarithm of the OPA titers and the corresponding CIs and based on the Student t distribution. Data for this outcome measure was planned to be analyzed for coadministration group (20vPnC + BNT162b2) and 20vPnC only group (20vPnC + saline) as specified in protocol.
Time Frame: 1 month after vaccination with 20vPnC
Population: Evaluable immunogenicity population (EIP): all randomized participants who received assigned vaccination; had at least 1 valid immunogenicity result from the blood sample collected within 20 to 49 days after vaccination at Day 1; had no other major protocol deviations as determined by clinician. Here, "Number Analyzed" signifies participants with valid OPA titers for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Coadministration Group: 20vPnC+BNT162b2 | 20vPnC Only Group: 20vPnC+Saline
Number analyzed (Participants) | 184 | 182
Titer
  Serotype 1: number analyzed (Participants) | 181 | 182
  Serotype 1 | 142 [116 to 176] | 131 [106 to 162]
  Serotype 3: number analyzed (Participants) | 180 | 182
  Serotype 3 | 49 [42 to 56] | 52 [44 to 61]
  Serotype 4: number analyzed (Participants) | 179 | 179
  Serotype 4 | 609 [484 to 766] | 573 [447 to 734]
  Serotype 5: number analyzed (Participants) | 179 | 179
  Serotype 5 | 81 [65 to 100] | 98 [80 to 120]
  Serotype 6A: number analyzed (Participants) | 182 | 181
  Serotype 6A | 1377 [1058 to 1792] | 1317 [1042 to 1665]
  Serotype 6B: number analyzed (Participants) | 180 | 182
  Serotype 6B | 1449 [1153 to 1821] | 1478 [1207 to 1810]
  Serotype 7F: number analyzed (Participants) | 182 | 182
  Serotype 7F | 977 [836 to 1142] | 1102 [951 to 1275]
  Serotype 8: number analyzed (Participants) | 175 | 179
  Serotype 8 | 299 [235 to 381] | 344 [274 to 431]
  Serotype 9V: number analyzed (Participants) | 180 | 179
  Serotype 9V | 1722 [1365 to 2172] | 1531 [1210 to 1936]
  Serotype 10A: number analyzed (Participants) | 179 | 177
  Serotype 10A | 2252 [1751 to 2898] | 2644 [2023 to 3456]
  Serotype 11A: number analyzed (Participants) | 170 | 165
  Serotype 11A | 1875 [1414 to 2488] | 1932 [1445 to 2583]
  Serotype 12F: number analyzed (Participants) | 177 | 169
  Serotype 12F | 2165 [1668 to 2809] | 2211 [1695 to 2885]
  Serotype 14: number analyzed (Participants) | 181 | 179
  Serotype 14 | 709 [572 to 879] | 640 [528 to 775]
  Serotype 15B: number analyzed (Participants) | 175 | 179
  Serotype 15B | 1520 [1092 to 2117] | 1852 [1377 to 2491]
  Serotype 18C: number analyzed (Participants) | 182 | 178
  Serotype 18C | 1059 [869 to 1290] | 846 [684 to 1046]
  Serotype 19A: number analyzed (Participants) | 181 | 179
  Serotype 19A | 637 [520 to 781] | 530 [436 to 644]
  Serotype 19F: number analyzed (Participants) | 181 | 182
  Serotype 19F | 305 [242 to 383] | 377 [299 to 476]
  Serotype 22F: number analyzed (Participants) | 168 | 167
  Serotype 22F | 5225 [3931 to 6943] | 4464 [3354 to 5942]
  Serotype 23F: number analyzed (Participants) | 182 | 182
  Serotype 23F | 336 [251 to 450] | 385 [283 to 524]
  Serotype 33F: number analyzed (Participants) | 170 | 172
  Serotype 33F | 4907 [3813 to 6316] | 5544 [4234 to 7261]

6. Secondary Outcome: Geometric Mean Concentration (GMC) of Full-Length S-Binding Immunoglobulin G (IgG) Levels at 1 Month After Vaccination With BNT162b2
Description: IgG levels were measured in serum samples using severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) full-length S-binding assay. GMCs and 2-sided CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs and based on the Student t distribution. Data for this outcome measure was planned to be analyzed for coadministration group (20vPnC + BNT162b2) and BNT162b2 only group (BNT162b2 + saline) as specified in protocol.
Time Frame: 1 month after vaccination with BNT162b2
Population: EIP: all randomized participants who received assigned vaccination; had at least 1 valid immunogenicity result from blood sample collected within 20 to 49 days after vaccination at Day 1; had no other major protocol deviations as determined by clinician. Participants with SARS-CoV-2 infection up to 1 month after vaccination (including subclinical infection, ie positive for N-binding antibody) were excluded from analysis. N=participants with valid assay results at specified sampling time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Units per milliliter
Arm/Group | Coadministration Group: 20vPnC+BNT162b2 | BNT162b2 Only Group: BNT162b2+Saline
Number analyzed (Participants) | 178 | 177
Units per milliliter | 29114 [26120 to 32451] | 26655 [24003 to 29599]

7. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Full-Length S-Binding IgG Levels From Before Vaccination to 1 Month After Vaccination With BNT162b2
Description: The GMFR for each vaccine group was defined as the geometric mean of the fold rises in the assay results from before to approximately 1 month after vaccination. GMFRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs and based on the Student t distribution. Data for this outcome measure was planned to be analyzed for coadministration group (20vPnC + BNT162b2) and BNT162b2 only group (BNT162b2 + saline) as specified in the protocol.
Time Frame: Before vaccination to 1 month after vaccination with BNT162b2
Population: EIP: participants received assigned vaccination; at least 1 valid immunogenicity result from sample collected within 20 to 49 days after Day1 vaccination; no other major protocol deviations determined by clinician. Participants with SARS-CoV-2 infection upto 1 month after vaccination (including subclinical infection, ie positive for N-binding antibody)excluded from analysis. N=participants with valid full-length S-binding IgG from before and 1 month after BNT162b2 booster dose sample collection.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Coadministration Group: 20vPnC+BNT162b2 | BNT162b2 Only Group: BNT162b2+Saline
Number analyzed (Participants) | 178 | 177
Fold rise | 35.5 [30.9 to 40.7] | 39.0 [33.5 to 45.5]

ADVERSE EVENTS:
Time Frame: Systematic assessment: local reactions recorded within 10 days after vaccination, and systemic events recorded within 7 days after vaccination; Non-systematic assessment: SAEs recorded from day of vaccination (Day 1) up to 6 months after vaccination and other AEs recorded from Day 1 up to 1 month after vaccination
Description: Same event may appear as AE and SAE but what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study.
Arm/Group | Coadministration Group: 20vPnC+BNT162b2 | 20vPnC Only Group: 20vPnC+Saline | BNT162b2 Only Group: BNT162b2+Saline
All-Cause Mortality (participants affected / at risk) | 1/187 | 0/187 | 0/185
Serious Adverse Events (participants affected / at risk) | 1/187 | 2/187 | 5/185
Other Adverse Events (participants affected / at risk) | 157/187 | 137/187 | 149/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coadministration Group: 20vPnC+BNT162b2 (N=187) | 20vPnC Only Group: 20vPnC+Saline (N=187) | BNT162b2 Only Group: BNT162b2+Saline (N=185)
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Coadministration Group: 20vPnC+BNT162b2 (N=187) | 20vPnC Only Group: 20vPnC+Saline (N=187) | BNT162b2 Only Group: BNT162b2+Saline (N=185)
Chills (CHILLS) (General disorders) | 49 | 13 | 41
Fatigue (FATIGUE) (General disorders) | 100 | 67 | 101
Injection site erythema (REDNESS) (General disorders) | 26 | 15 | 22
Injection site pain (PAIN) (General disorders) | 146 | 115 | 133
Injection site swelling (SWELLING) (General disorders) | 26 | 16 | 21
Pyrexia (FEVER) (General disorders) | 24 | 2 | 16
Urinary tract infection (Infections and infestations) | 2 | 0 | 1
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 49 | 17 | 46
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 60 | 27 | 59
Dizziness (Nervous system disorders) | 2 | 0 | 0
Headache (HEADACHE) (Nervous system disorders) | 56 | 32 | 61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT04887948/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/48/NCT04887948/SAP_001.pdf